CLINICAL TRIAL: NCT00769132
Title: A Randomized, Double-Blind, Placebo-Controlled, 4-Period, Crossover Study to Evaluate the Effects of ER Niacin/Laropiprant, Laropiprant, ER Niacin, and Placebo on Urinary Prostanoid Metabolites in Subjects With Hypercholesterolemia
Brief Title: A Study to Evaluate the Effects of Extended Release (ER) Niacin/Laropiprant, Laropiprant, ER Niacin, and Placebo on Urinary Prostanoid Metabolites in Subjects With High Cholesterol (0524A-075)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-075; 2008_561
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2008-11-27 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — MK-0524; Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- A (Experimental): ER niacin/laropiprant + Placebo to laropiprant
  Interventions: Drug: Comparator: niacin + laropiprant
- B (Active Comparator): ER niacin + Placebo to laropiprant
  Interventions: Drug: Comparator: niacin
- C (Experimental): laropiprant + Placebo to ER niacin/laropiprant
  Interventions: Drug: Comparator: laropiprant
- D (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: Comparator: niacin + laropiprant — ER niacin 2 g/laropiprant 40 mg tablet once daily for 7 days
  Arms: A
Drug: Comparator: niacin — ER niacin 2 g tablet once daily for 7 days
  Other Names: Niaspan
  Arms: B
Drug: Comparator: laropiprant — laropiprant 40 mg once daily for 7 days
  Arms: C
Drug: Comparator: placebo — matching placebo tablets for each of the interventions once daily for 7 days
  Arms: D

SUMMARY:
The purpose of this study is to evaluate the potential effects of ER niacin/laropiprant, ER niacin, laropiprant, and placebo over the course of seven days on urinary levels of a metabolite of thromboxane A2 (TxA2), as a marker of in vivo platelet reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects may not be pregnant and/or will agree to use appropriate method of contraception beginning at least 2 weeks prior to administration of the first dose of study drug in the first treatment period, throughout the study and until at least 2 weeks after administration of the last dose of study drug in the last treatment period.
* Subject is judged to be in good health based on medical history, physical examination, vital sign measurements, and laboratory safety tests performed at the prestudy (screening) visit and/or prior to administration of the initial dose of study drug.
* Subject has no clinically significant abnormality on electrocardiogram (ECG) performed at the prestudy (screening) visit and/or prior to administration of the initial dose of study drug.
* Subject has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months; subjects who have discontinued smoking or the use of nicotine/nicotine containing products for at least approximately 3 months may be enrolled in the study at the discretion of the investigator

Exclusion Criteria:

* Subject is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder over the last 5 to 10 years. - Subjects who have had situational depression may be enrolled in the study at the discretion of the investigator.
* Subject has a history of stroke, chronic seizures, or major neurological disorder.
* Subject has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases.
* Subject has a history of neoplastic disease (including leukemia, lymphoma, malignant melanoma), or myeloproliferative disease, regardless of the time since treatment.
* Subject has history of a thrombotic or platelet related disorder including prior deep venous thrombosis. Subject is being treated with coumadin, heparin, clopidogrel has used these agents within 2 weeks of screening. Subject is being treated with aspirin or has used this agent within 3 weeks prior to administration of screening.
* Subject is unable to refrain from or anticipates the use of any medication, including prescription and non- prescription drugs or herbal remedies beginning approximately 2 weeks prior to administration of the initial dose of study drug, throughout the study until the poststudy visit.
* Subject consumes excessive amounts of alcohol, defined as greater than 3 glasses, of alcoholic beverages or distilled spirits per day.
* Subject consumes excessive amounts, defined as greater than 6 servings, of coffee, tea, cola, or other caffeinated beverages per day.
* Subject has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks prior to the prestudy (screening) visit.
* Subject has a history of significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food.
* Subject is currently a regular user of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-08-03 (Actual); Primary Completion 2007-10-13 (Actual); Study Completion 2007-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lauring B, Dishy V, Luo WL, Laterza O, Patterson J, Cote J, Chao A, Larson P, Gutierrez M, Wagner JA, Lai E. Laropiprant in combination with extended-release niacin does not alter urine 11-dehydrothromboxane B2, a marker of in vivo platelet function, in healthy, hypercholesterolemic, and diabetic subjects. J Clin Pharmacol. 2009 Dec;49(12):1426-35. doi: 10.1177/0091270009339593. Epub 2009 Oct 15. PMID 19833861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I
  First Patient Entered 16 Aug 2007.
  Study conducted at Comprehensive Phase One, Miramar, FL. and Cedra Clinical Research LLC, San Antonio, TX.
Groups:
- Sequence 1: D/C/A/B: A = Extended Release (ER) niacin 2 g/laropiprant 40 mg once daily for 7 days
  B = ER niacin 2 g once daily for 7 days
  C = laropiprant 40 mg once daily for 7 days
  D = placebo once daily for 7 days
- Sequence 2: C/B/D/A; Sequence 3: B/A/C/D; Sequence 4: A/D/B/C: A = ER niacin 2 g/laropiprant 40 mg once daily for 7 days B = ER niacin 2 g once daily for 7 days
  C = laropiprant 40 mg once daily for 7 days
  D = placebo once daily for 7 days
Period: Period 1
Arm/Group | Sequence 1: D/C/A/B | Sequence 2: C/B/D/A | Sequence 3: B/A/C/D | Sequence 4: A/D/B/C
Started | 7 | 6 | 6 | 7
Completed | 6 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 1
Period: Period 2
Arm/Group | Sequence 1: D/C/A/B | Sequence 2: C/B/D/A | Sequence 3: B/A/C/D | Sequence 4: A/D/B/C
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Period 3
Arm/Group | Sequence 1: D/C/A/B | Sequence 2: C/B/D/A | Sequence 3: B/A/C/D | Sequence 4: A/D/B/C
Started | 6 | 6 | 6 | 5
Completed | 5 | 6 | 6 | 5
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1: D/C/A/B | Sequence 2: C/B/D/A | Sequence 3: B/A/C/D | Sequence 4: A/D/B/C
Started | 5 | 6 | 6 | 5
Completed | 5 | 5 | 6 | 5
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Totals for Study: All participants in the study.
Arm/Group | Totals for Study
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (11.6) [22 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Height [Mean (Full Range); unit: cm] | 165.5 [147.0 to 185.0]
Weight [Mean (Full Range); unit: kg] | 78.4 [58.0 to 102.9]
urinary 11-dTxB2 [Median (Full Range); unit: pg/mg creatinine] — urinary levels of 11-dehydrothromboxane B2 (24 hour collection)
  pg/mg creatinine | 418.5 [142.0 to 783.1]
urinary PGI2-Metabolite [Median (Full Range); unit: pg/mg creatinine] — urinary levels of 2,3-dinor 6-keto-PGF1a (Prostaglandin I-M) 24-hour collection
  pg/mg creatinine | 89.7 [45.2 to 242.9]

OUTCOME MEASURES:

1. Primary Outcome: Urinary 11-dehydrothromboxane B2 (11-dTxB2)
Description: The creatinine-normalized urine levels of 11-dTxB2 on Day 7 following a 7 day course of daily dosing in the overall 24 hour collection interval.
Time Frame: On Day 7 across the 24-hour urinary collection period.
Population: Twenty-six (26) subjects (including replacements) were enrolled in this study. All available subjects (besides the 4 that were excluded due suspected NSAID/Aspirin use) and had partial data (at least one available period) were included in the statistical analysis models/comparisons.
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mg creatinine
Groups:
- ER Niacin 2 g / Laropiprant 40 mg: ER niacin 2 g/laropiprant 40 mg daily for 7 days
- ER Niacin 2 g: ER niacin 2 g daily for 7 days
- Laropiprant 40 mg: Laropiprant 40 mg once daily for 7 days
- Placebo: Placebo daily for 7 days
Arm/Group | ER Niacin 2 g / Laropiprant 40 mg | ER Niacin 2 g | Laropiprant 40 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 19 | 20
pg/mg creatinine | 414.6 [316.8 to 542.6] | 371.6 [283.8 to 486.5] | 407.3 [312.2 to 531.4] | 466.1 [358.4 to 606.3]
Statistical Analysis 1: Comparison: ER Niacin 2 g / Laropiprant 40 mg vs ER Niacin 2 g; The endpoint is the urine levels of 11-dTxB2 on Day 7 following a 7 day course of daily dosing in the overall 24 hour collection interval. The point estimate and 90% confidence intervals (CIs) were calculated for the geometric mean ratio (GMR) [Treatment A/B] of the urine levels of 11-dTxB2 on Day 7; Test type: Non-Inferiority or Equivalence — Two treatments are comparable if the geometric mean ratio is contained within the interval [0.50-2.00]; Geometric least-squares mean ratio = 1.12, 90% CI [0.9 to 1.38]
Statistical Analysis 2: Comparison: Laropiprant 40 mg vs Placebo; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.87, 90% CI [0.71 to 1.07]
Statistical Analysis 3: Comparison: ER Niacin 2 g vs Placebo; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.8, 90% CI [0.65 to 0.98]
Statistical Analysis 4: Comparison: ER Niacin 2 g / Laropiprant 40 mg vs Placebo; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.89, 90% CI [0.72 to 1.09]
Statistical Analysis 5: Comparison: ER Niacin 2 g vs Laropiprant 40 mg; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.91, 90% CI [0.74 to 1.12]
Statistical Analysis 6: Comparison: ER Niacin 2 g / Laropiprant 40 mg vs Laropiprant 40 mg; Test type: Superiority or Other; Geometric least-squares mean ratio = 1.02, 90% CI [0.83 to 1.25]

2. Secondary Outcome: Prostaglandin I Metabolite (PGI-M)
Description: The creatinine-normalized urine levels of PGI-M in the overall 24 hour collection interval following administration on Day 7.
Time Frame: On Day 7 across the 24-hour urinary collection period.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mg creatinine
Arm/Group | ER Niacin 2 g / Laropiprant 40 mg | ER Niacin 2 g | Laropiprant 40 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 19 | 20
pg/mg creatinine | 73.5 [61.4 to 88.1] | 70.9 [59.2 to 85.0] | 114.5 [95.6 to 137.2] | 127.5 [106.6 to 152.4]
Statistical Analysis 1: Comparison: ER Niacin 2 g / Laropiprant 40 mg vs ER Niacin 2 g; Test type: Superiority or Other; Geometric least-squares mean ratio = 1.04, 90% CI [0.92 to 1.17]
Statistical Analysis 2: Comparison: Laropiprant 40 mg vs Placebo; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.9, 90% CI [0.8 to 1.01]
Statistical Analysis 3: Comparison: ER Niacin 2 g vs Placebo; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.56, 90% CI [0.49 to 0.63]
Statistical Analysis 4: Comparison: ER Niacin 2 g / Laropiprant 40 mg vs Placebo; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.58, 90% CI [0.51 to 0.65]
Statistical Analysis 5: Comparison: ER Niacin 2 g vs Laropiprant 40 mg; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.62, 90% CI [0.55 to 0.7]
Statistical Analysis 6: Comparison: ER Niacin 2 g / Laropiprant 40 mg vs Laropiprant 40 mg; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.64, 90% CI [0.57 to 0.72]

ADVERSE EVENTS:
Description: Although 26 participants were included in the assessment of safety, not all participants received all treatments.
Groups:
- ER Niacin 2 g / Laropiprant 40 mg: ER niacin 2 g/laropiprant 40 mg once daily for 7 days
- ER Niacin 2 g: ER niacin 2 g once daily for 7 days
- Placebo: Placebo once daily for 7 days
Arm/Group | ER Niacin 2 g / Laropiprant 40 mg | ER Niacin 2 g | Laropiprant 40 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 15/25 | 21/24 | 4/25 | 5/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ER Niacin 2 g / Laropiprant 40 mg (N=25) | ER Niacin 2 g (N=24) | Laropiprant 40 mg (N=25) | Placebo (N=25)
Gastrointestinal Disorders (Gastrointestinal disorders) | 7 | 7 | 3 | 3
Abdominal Pain (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 1
Dry Mouth (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 3 | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3 | 2 | 0
General Disorders And Administration Site Conditions (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Musculoskeletal And Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Nervous System Disorders (Nervous system disorders) | 8 | 5 | 2 | 3
Headache (Nervous system disorders) | 7 | 4 | 1 | 3
Renal And Urinary Disorders (Renal and urinary disorders) | 0 | 0 | 1 | 2
Skin And Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 2 | 5 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5 | 1 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Vascular Disorders (Vascular disorders) | 8 | 20 | 2 | 1
Flushing (Vascular disorders) | 8 | 20 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.